CLINICAL TRIAL: NCT01139931
Title: Epigenetic Alterations in AML
Brief Title: Biomarker Changes in Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B9; COG-AAML10B9 (Other: Children's Oncology Group); CDR0000671474 (Other: Clinical Trials.gov); NCI-2011-02225 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood or tumor tissue from patients with cancer in the laboratory may help doctors learn about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarker changes in samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Map key histone modifications and cytosine methylation in leukemia cell lines with defined oncogenic mutations.
* Acquire genome-wide maps of key histone modifications and cytosine methylation for primary leukemia in samples from patients with acute myeloid leukemia (AML).
* Investigate functional relationships between genetic and epigenetic landscapes in AML.

OUTLINE: Archived samples are analyzed in vivo and in vitro (cell line) for histone modification and cytosine methylation. Genome-wide locations of 5 histone modifications are analyzed using chip-Seq, as well as DNA methylation analysis at nucleotide-resolution by high-throughput bisulfite sequencing. These epigenetic data are correlated with genomic data (sequence analysis, expression array, SNP array).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Primary leukemia samples from the Children Oncology Group (COG) bank with sufficient number of cells (500,000-1 million cells) with > 80% of leukemia blasts

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Diagnosis of acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Relationships between genetic and epigenetic landscapes in AML

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Fred Hutchinson Cancer Center